CLINICAL TRIAL: NCT07351565
Title: Chemotherapy Plus Pitavastatin Guided by Patient-Derived Tumor-like Cell Clusters in Refractory Non-Small Cell Lung Cancer: An Exploratory Phase I Trial
Brief Title: Chemotherapy Plus Pitavastatin Guided by Patient-Derived Tumor-like Cell Clusters in Refractory Non-Small Cell Lung Cancer
Acronym: CPPGPTCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chang Chen (Other)
Responsible Party: Sponsor-Investigator, Chang Chen, director of hospital, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L25-751-1
Record Dates: First submitted 2025-12-27; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pitavastatin plus chemotherapy (Experimental): The drugs used in this arm included chemotherapy agents such as cisplatin for injection, carboplatin for injection, pemetrexed disodium for injection, paclitaxel injection, gemcitabine hydrochloride for injection, and docetaxel injection, as well as pitavastatin. Treatment plan: The selection of chemotherapy drugs was based on the results of PTC drug sensitivity testing, with combination therapy showing the highest sensitivity. Drug dosages were administered according to the recommended standards outlined in the guidelines (every three weeks, intravenous). Treatment continued until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of treatment for other reasons specified in the protocol, whichever occurred first. Pitavastatin is administered orally by the subjects themselves at a fixed time each morning (4 mg, once daily), with or without food, until disease progression or intolerance occurs.
  Interventions: Drug: Pitavastatin 1 mg daily or 4 mg daily

INTERVENTIONS:
Drug: Pitavastatin 1 mg daily or 4 mg daily — The selection of chemotherapy drugs was based on the results of PTC drug sensitivity testing, with combination therapy showing the highest sensitivity. Drug dosages were administered according to the recommended standards outlined in the guidelines (every three weeks, intravenous). Treatment continued until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of treatment for other reasons specified in the protocol, whichever occurred first.
  Pirvastatin is administered orally by the subjects themselves at a fixed time each morning (4 mg, once daily), with or without food, until disease progression or intolerance occurs.

SUMMARY:
The primary objective of this study is to evaluate the objective response rate (ORR = CR + PR) of pitavastatin combined with chemotherapy, guided by PTC (patient-derived tumor-like cell cluster) drug sensitivity, in patients resistant to second-line treatment (PD/SD). The ORR is defined as the proportion of patients achieving a response after four cycles of combination therapy. The main questions it aims to answer are:

1. Does PTC-guided medication is feasible
2. Does the administration of Pitavastatin combined with chemotherapy can improve the objective response rate (ORR) in second-line drug-resistant patients

The medication to participants will be strictly guided by PTC drug testing. The drugs examined in this study included chemotherapy agents such as cisplatin for injection, carboplatin for injection, pemetrexed disodium for injection, paclitaxel injection, gemcitabine hydrochloride for injection, and docetaxel injection, as well as pitavastatin. The selection of chemotherapy drugs was based on the results of PTC drug sensitivity testing, with combination therapy showing the highest sensitivity. Drug dosages were administered according to the recommended standards outlined in the guidelines (every three weeks, intravenous). Treatment continued until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of treatment for other reasons specified in the protocol, whichever occurred first.

Pirvastatin is administered orally by the subjects themselves at a fixed time each morning (4 mg, once daily), with or without food, until disease progression or intolerance occurs. Participants must demonstrate good compliance throughout the entire study, especially when the dosage is reduced, to ensure they receive the correct prescribed dose.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years old.
* Non-small cell lung cancer diagnosed through pathological methods (including histology or cytology).
* Resistance to second-line drug therapy, with imaging (based on RECIST 1.1 criteria) confirming tumor response as either progressive disease (PD) or stable disease (SD).
* Presence of measurable lesions according to RECIST 1.1 criteria: tumor lesions must have a CT scan length of ≥ 10 mm; lymph node lesions must have a CT scan short diameter of ≥ 15 mm; scan slice thickness should not exceed 5 mm; and measurable lesions must not have undergone local treatments such as radiotherapy or cryotherapy.
* ECOG Performance Status: 0-2 points.
* Expected survival period of at least 6 months.
* Hematological function is considered sufficient, defined as: absolute neutrophil count ≥ 1.5 × 10^9/L; platelet count ≥ 80 × 10^9/L; hemoglobin ≥ 90 g/L (no history of blood transfusion within the past 7 days, and not corrected with G-CSF or other hematopoietic stimulating factors).
* Adequate liver function defined as having total bilirubin levels ≤ 1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times the ULN.
* Adequate renal function, defined as a creatinine clearance rate of ≥ 50 mL/min (calculated using the Cockcroft-Gault formula).
* Adequate coagulation function defined as an International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times the upper limit of normal (ULN). If the subject is receiving anticoagulant therapy, coagulation function is considered adequate as long as the INR/PT values fall within the therapeutic range specified for the anticoagulant medication.
* For female subjects of childbearing age, a negative urine or serum pregnancy test must be conducted within three days prior to the first administration of the study drug. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required.
* If there is a risk of conception, male and female patients should use highly effective contraception (i.e., methods with an annual failure rate of less than 1%) and continue for at least 180 days after stopping the trial treatment. Note: If abstinence is the subject's usual lifestyle and preferred contraceptive method, then abstinence is acceptable.
* The subjects voluntarily joined this study, signed a written informed consent form before any trial-related procedures were implemented, demonstrated good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Individuals known to be allergic to the active or inactive ingredients of pitavastatin, or to drugs with chemical structures similar to pitavastatin.
* Individuals with known allergies to pemetrexed, paclitaxel, gemcitabine, or platinum.
* Active hemoptysis, active diverticulitis, abdominal abscess, and gastrointestinal obstruction requiring clinical intervention.
* Symptomatic, uncontrolled brain metastases or leptomeningeal metastases, or controlled brain metastases with symptoms lasting less than 2 months.
* Diagnosed with malignant tumors other than small cell lung cancer within two years prior to enrollment, excluding completely treated basal or squamous cell skin cancer and/or radically resected in situ cancer.
* Has undergone major surgery within the 4 weeks prior to the start of the study or has experienced complications or sequelae that have not yet resolved.
* Suffering from serious or uncontrolled illnesses, including but not limited to: uncontrollable nausea and vomiting; inability to alleviate symptoms of intestinal obstruction; inability to swallow study medications; gastrointestinal diseases that may interfere with drug absorption and metabolism; respiratory syndrome caused by pleural effusion or ascites (≥ CTCAE grade 2 dyspnea); active viral infections (HIV, HBV, HCV); or uncontrolled epileptic seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental disorders hindering informed consent.
* Having a tendency to bleed and a history of thrombosis, specifically:
* Any bleeding events of CTCAE grade 2 occurring within the first 3 months of screening, or grade 3 or higher within the first 6 months.
* Active bleeding, coagulation dysfunction, bleeding tendency, or current treatment with thrombolytic or anticoagulant therapy.
* Requirement for anticoagulant therapy with medications such as warfarin or heparin.
* Requirement for long-term antiplatelet therapy, such as aspirin or clopidogrel.
* Thrombotic or embolic events within the past six months (including CVA/TIA and pulmonary embolism).
* Significant cardiovascular history, specifically:
* NYHA Class III and IV congestive heart failure.
* Unstable angina, newly diagnosed angina, or myocardial infarction within the previous 12 months.
* Arrhythmia requiring therapeutic intervention (patients taking beta blockers or digoxin may be enrolled).
* CTCAE Grade ≥ 2 valvular heart disease.
* Poor control of hypertension (systolic BP > 150 mmHg or diastolic BP > 100 mmHg).
* History of non-infectious pneumonia requiring corticosteroid treatment within one year prior to enrollment, or a current diagnosis of non-infectious pneumonia.
* Any past or current diseases, treatments, or laboratory abnormalities that may interfere with the research results, affect the patient's full participation, or lead the researcher to believe that the patient is unsuitable to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the date of first dose until disease progression or death from any cause, assessed up to 6 months.
  ORR is defined as the proportion of participants with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) according to RECIST v1.1.

IPD SHARING:
Plan to Share IPD: Undecided